CLINICAL TRIAL: NCT07031414
Title: Comparison of Ultrasonography-Guided Residual Gastric Volume Measurement Before Elective Surgery in Diabetic and Non-Diabetic Patients
Brief Title: Preoperative Residual Gastric Volume
Status: Active, not recruiting | Type: Observational
Sponsor: Izmir City Hospital (Other Government)
Responsible Party: Principal Investigator, Derya Arslan Yurtlu, Professor, Izmir City Hospital
Other Study IDs: IZMIR CITY HOSPİTAL; IZMIR CITY HOSPİTAL (Other: IZMIR CITY HOSPİTAL)
Record Dates: First submitted 2025-06-12; First posted 2025-06-22 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Preoperative; Gastric; Residual Volume
Keywords: Ultrasonography-Guided; Residual gastric volume; Diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Biospecimen Retention: Samples Without DNA — No specimen
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Diabetic Group - Patients with a diagnosis of diabetes mellitus Non-Diabetic Group - Patients witho: Diabetic Group Adult patients (aged 18-65) with a known diagnosis of diabetes mellitus who are scheduled for elective surgery under general anesthesia.
  These participants will undergo preoperative bedside gastric ultrasound to evaluate residual gastric volume, content type, and aspiration risk.
  Non-Diabetic Group Adult patients (aged 18-65) without diabetes mellitus, scheduled for elective surgery under general anesthesia.
  These participants will also undergo preoperative bedside gastric ultrasound for the same assessments as the diabetic group.

SUMMARY:
The goal of this observational study is to assess the preoperative gastric residual volume in adult patients undergoing elective surgery. The main question it aims to answer is:

Does gastric residual volume, content type, and aspiration risk differ between diabetic and non-diabetic patients with similar fasting durations?

Participants undergoing elective surgery will receive bedside gastric ultrasound as part of their preoperative assessment. Ultrasound images will be used to estimate gastric volume and evaluate aspiration risk.

DETAILED DESCRIPTION:
The goal of this observational study is to assess whether bedside gastric ultrasound can identify differences in residual gastric volume, content type, and aspiration risk in adult diabetic and non-diabetic patients (ages 18-65) undergoing elective surgery under general anesthesia.

The main questions it aims to answer are:

Do diabetic patients have higher residual gastric volume than non-diabetic patients despite similar fasting durations?

Does the type or amount of gastric content differ between the two groups, potentially increasing aspiration risk?

Researchers will compare diabetic and non-diabetic groups to see if diabetes is associated with delayed gastric emptying and increased aspiration risk.

Participants will:

Undergo bedside gastric ultrasound prior to anesthesia induction

Be scanned in semi-sitting and right lateral decubitus positions using a convex ultrasound probe

Have gastric antrum graded and volume calculated

Be evaluated for aspiration risk based on validated ultrasound criteria

ELIGIBILITY:
Inclusion Criteria:Male and female patients

* Aged 18 to 65 years,
* American Society of Anesthesiologists (ASA) physical status I -III
* Scheduled for elective surgery under general anesthesia.
* Patients with a known history of diabetes mellitus will be included in the diabetic group.

Exclusion Criteria:Male and female patients

* Pregnant patients
* Patients with gastrointestinal obstructive diseases
* Patients with gastroesophageal reflux disease
* History of gastrointestinal surgery
* Emergency surgery cases
* Recent history of abdominal trauma
* Non-diabetic patients with autonomic or neurological disorders
* Patients with chronic kidney disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of adult patients aged 18 to 65 years, of both sexes, who are scheduled for elective surgery under general anesthesia. Participants will be classified into two groups: those with a documented history of diabetes mellitus (diabetic group) and those without (non-diabetic group). All patients will have American Society of Anesthesiologists (ASA) physical status I-III. The study will be conducted at Izmir City Hospital, and only patients who provide written informed consent will be included.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2025-03-15 (Actual); Primary Completion 2025-08-15 (Estimated); Study Completion 2025-08-15 (Estimated)

PRIMARY OUTCOMES:
Residual gastric volume (mL) measured by bedside ultrasound in diabetic vs. non-diabetic patients. | Immediately before induction of anesthesia (preoperative period)
  The main question of the study is whether gastric emptying is delayed in diabetic patients, resulting in a higher residual gastric volume.

CONTACTS AND LOCATIONS:
Overall Officials: Derya A. Yurtlu, M.D., Principal Investigator — Izmir City Hospital, Izmir, TURKEY
Locations (1):
- University of Health Sciences, Izmir Faculty of Medicine, Izmir City Hospital, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The reason is that the local health authority (Provincial Health Directorate) did not grant permission for the sharing of individual participant-level data with external researchers.